CLINICAL TRIAL: NCT00804193
Title: A Double-blind, Randomized, Parallel-group, Vehicle-controlled, Multi-center Study to Evaluate the Safety and Clinical Equivalence of a Generic Ciclopirox Olamine Topical Suspension to Reference Ciclopirox Topical Suspension 0.77% in the Treatment of Tinea Pedis
Brief Title: Safety and Equivalence of a Generic Ciclopirox Olamine Topical Suspension Compared to the Reference Ciclopirox Topical Suspension 0.77% for the Treatment of Tinea Pedis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPL-402
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Tinea Pedis
Keywords: Tinea Pedis; Ciclopirox Olamine
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test Product (Experimental): Ciclopirox Olamine Topical Suspension
  Interventions: Drug: Ciclopirox Olamine Topical Suspension
- Reference Product (Active Comparator): Loprox® Topical Suspension 0.77%
  Interventions: Drug: Ciclopirox Topical Suspension 0.77%-Reference Product
- Vehicle Product (Placebo Comparator): placebo of test product
  Interventions: Drug: Ciclopirox Olamine Topical Suspension-Placebo

INTERVENTIONS:
Drug: Ciclopirox Olamine Topical Suspension — topical suspension
  Arms: Test Product
Drug: Ciclopirox Topical Suspension 0.77%-Reference Product — topical suspension
  Arms: Reference Product
Drug: Ciclopirox Olamine Topical Suspension-Placebo — topical suspension
  Arms: Vehicle Product

SUMMARY:
The objectives of this study were to demonstrate comparable safety and efficacy of Ciclopirox Olamine Topical Suspension (Test Product) and Ciclopirox Topical Suspension 0.77% (Reference Product) in the treatment of subjects with tinea pedis, and to show the superiority of the active treatments over that of the vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 10 years of age, and otherwise healthy
* Clinically and mycologically confirmed diagnosis of symptomatic tinea pedis
* In good health with no clinically significant disease that might have interfered with study evaluations
* Study participant or legal guardian was willing and able to read and sign an IRB approved ICF, which included agreement to comply with all study requirements as indicated in the protocol. For subjects 10 to 17 years of age, an assent form for minors was completed.

Exclusion Criteria:

* History of hypersensitivity or allergy to ciclopirox
* Had any skin condition that would interfere with the diagnosis or assessment of tinea pedis
* Had a history of dermatophyte infection unresponsive to antifungal treatment
* Had a history of alcoholism, drug abuse, or problems that would likely have made the subject unreliable for the study
* Had any condition or used any medication that, in the opinion of the Investigator, might have interfered with the conduct or results of the study or placed the prospective subject at increased risk
* Was unwilling to sign the informed consent
* Female who was pregnant or lactating

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2004-06; Primary Completion 2004-12 (Actual); Study Completion 2005-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product: Ciclopirox Olamine Topical Suspension; the Test Product was applied treatment two times a day for 4 weeks
- Reference Product: Loprox® Topical Suspension 0.77%; the Reference Product was applied treatment two times a day for 4 weeks
- Vehicle Product: placebo of test product was applied treatment two times a day for 4 weeks
Period: Overall Study
Arm/Group | Test Product | Reference Product | Vehicle Product
Started | 220 | 224 | 109
Completed | 181 | 180 | 77
Not Completed | 39 | 44 | 32
Not completed — Lack of baseline fungus | 32 | 31 | 19
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Lack of Efficacy | 1 | 1 | 3
Not completed — Protocol Violation | 0 | 8 | 2
Not completed — Lost to Follow-up | 3 | 3 | 4
Not completed — Withdrawal by Subject | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference Product | Vehicle Product | Total
Number analyzed (Participants) | 220 | 224 | 109 | 553
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 13 | 4 | 27
  Between 18 and 65 years | 188 | 181 | 86 | 455
  >=65 years | 22 | 30 | 19 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (16.0) | 44.1 (16.5) | 47.7 (16.5) | 45.1 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 68 | 33 | 166
  Male | 155 | 156 | 76 | 387
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 60 | 26 | 141
  Not Hispanic or Latino | 165 | 164 | 83 | 412
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 2 | 5 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 37 | 26 | 21 | 84
  White | 178 | 192 | 82 | 452
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 220 | 224 | 109 | 553

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects in Each Treatment Group With Therapeutic Success
Description: Therapeutic success was defined as having both Mycological Cure (potassium hydroxide [KOH] wet mount negative and fungal culture negative) and Clinical Cure
Time Frame: 6 weeks
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | Test Product | Reference Product | Vehicle Product
Number analyzed (Participants) | 149 | 165 | 74
participants | 93 | 88 | 7
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — 90% CI was constructed for the difference in the Therapeutic Success rates between the Test Product and Reference Product at Visit 4/Week 6 (Follow-Up). The interval was calculated using Wald's method with Yates' continuity correction. Therapeutic equivalence (bioequivalence) was established if this 90% CI was contained within the interval -0.20 to +0.20 (-20% to +20%); Wald's method, Yates; CI calculated using Wald's method with Yates' continuity correction; Difference in Percentage of Participants = 9, 90% CI 2-sided [-0.69 to 18.85] — The sample size for this study was calculated assuming that both active treatments would have equivalent success proportions of at least 55% and the Vehicle would have a success proportion no greater than 25%

2. Secondary Outcome: Proportion of Subjects With Mycological Cure
Description: Potassium hydroxide [KOH] wet mount negative and fungal culture negative
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Test Product | Reference Product | Vehicle Product
Number analyzed (Participants) | 149 | 165 | 74
participants | 119 | 127 | 18
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — 90% CI was constructed for the difference in the Success rates between the Test Product and Reference Product at Visit 4/Week 6 (Follow-Up). The interval was calculated using Wald's method with Yates' continuity correction. Bioequivalence was established if this 90% confidence interval was contained within the interval -0.20 to +0.20); p = 0.001, Wald's method with Yates' continuity cor; Difference in Percentage of Participants = 1, 90% CI 2-sided [-7.08 to 9.24] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Proportion of Subjects With Clinical Cure
Description: Clinical Cure was defined as a signs and symptoms score of <1 for erythema; <1 for scaling; and 0 for pruritus, maceration, fissuring/cracking, and burning/stinging; as well as an assessment that no additional antifungal therapy was required to treat the subject's current episode of tinea pedis
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Test Product | Reference Product | Vehicle Product
Number analyzed (Participants) | 149 | 165 | 74
participants | 81 | 96 | 22
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.001, Wald's method Yates' continuity cor; Difference in Percentage of Participants = 4, 90% CI 2-sided [-4.60 to 14.24] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Test Product | Reference Product | Vehicle Product
Serious Adverse Events (participants affected / at risk) | 0/220 | 2/224 | 4/109
Other Adverse Events (participants affected / at risk) | 0/220 | 0/224 | 0/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=220) | Reference Product (N=224) | Vehicle Product (N=109)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Perforated sigmoid colon (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid hemorrhage; MCA aneurysm; PCOM (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Blood clots spleen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Seizures (transient ischaemic attack) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Right hip fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other